CLINICAL TRIAL: NCT06321367
Title: Construction and Validation of a Predictive Model of Coinfections in Elderly COVID-19 Patients After Abandoning Zero Policy
Brief Title: Model to Predict Coinfection in Elderly Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202401002; 82070613 (Other Grant/Funding Number: the National Natural Sciences Foundation of China); 82370638 (Other Grant/Funding Number: the National Natural Sciences Foundation of China); 2022RC1212 (Other Grant/Funding Number: the Science and Technology Innovation Program of Hunan Province); 2023JJ10095 (Other Grant/Funding Number: he Natural Science Foundation of Hunan Province China)
Record Dates: First submitted 2024-03-19; First posted 2024-03-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Covid19
Keywords: COVID-19; elderly; nomogram; coinfections; diagnosis
MeSH Terms: conditions — COVID-19; Coinfection; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- elderly COVID-19 patients with coinfection
- elderly COVID-19 without coinfection

SUMMARY:
The goal of this observational study is to learn about the clinical characteristics and construction of a predictive model in elderly COVID-19 patients. The main question it aims to answer is the main clinical characteristics and risk factors of elderly COVID-19 patients. Participants will not be asked to do any other intervening measure.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65 years old;
* COVID-19 was diagnosed with SARS-CoV-2 reverse transcription-polymerase chain reaction positive or rapid antigen test positive or a clinical diagnosis made by the radiological responsible clinician based on signs, symptoms, or radiology consistent with COVID-19;
* Hospitalization more than one day, including patients in emergency.

Exclusion Criteria:

* Age less than 65 years old;
* Pregnancy;
* Hospitalization less than one day;
* Outpatients;
* Patients with missing or incomplete information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly COVID-19 patients admitted into Xiangya Hospital of Central South University (in Changsha, Hunan) and Xiangya Hospital of Central South University, Jiangxi (in Nanchang, Jiangxi)
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Coinfection | from admission to 7 days after admission
  The investigators defined coinfection as coinfected bacteria, fungi, or other viruses with SARS-CoV-2 that occurred from admission to 7 days after admission. If a diagnosis was at the time of or within the first 48 hours of COVID-19 hospital admission, these infections were defined as community-acquired infections. If diagnosis occurred ≥48 hours to 7 days after admission for COVID-19, these infections were defined as early-onset hospital-acquired infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No